CLINICAL TRIAL: NCT05633719
Title: Multicenter, Prospective Observational Study for Early Diagnosis, and Development of Follow-up Protocol and Hearing Rehabilitation Program for Ototoxic Hearing Loss After Chemotherapy for Pediatric Solid Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Moo Kyun, Park, Professor, Seoul National University Hospital
Other Study IDs: 2208-162-1354
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumor, Childhood
Keywords: Pediatric solid tumor, Chemotherapy, Hearing loss
MeSH Terms: conditions — Hearing Loss | interventions — Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric solid cancer
  Interventions: Other: Chemotherapy involving cisplatin or carboplatin

INTERVENTIONS:
Other: Chemotherapy involving cisplatin or carboplatin — Chemotherapy

SUMMARY:
More than half of all pediatric cancer in Korea are solid cancer. For the treatment of solid cancer, multidisciplinary methods such as surgery, chemotherapy, and radiation therapy are applied, and with the development of the treatment method, the treatment performance has improved dramatically, and the 5-year survival rate of more than 80% is currently recorded. Due to the improvement in survival rate, interest in side effects caused by cancer treatment itself is gradually increasing, and efforts to reduce them are increasing. Accordingly, it aims to contribute to improving the quality of life of pediatric solid cancer survivors. by developing a Korean-type early diagnosis and follow-up protocol of ototoxic hearing loss, which commonly occurs in pediatric solid cancer who have undergone chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

① Solid cancer patients under the age of 19 receiving Platinum chemotherapy

② Solid cancer patients under the age of 19 receiving 30 Gy or more head and neck radiation therapy

Exclusion Criteria:

① Those who have received chemotherapy or radiation in the past

* Those who have difficulty understanding the clinical trial due to mental retardation or unable to read the consent form, such as illiteracy or foreigners ③ Those who have difficulty in hearing test due to neurological factors, etc. ④ Other cases judged to be inappropriate for this study by the judgment of the person in charge of the clinical trial

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are diagnosed as solid cancer and receive platinum chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ototoxic hearing loss | 1 year after the initiation of chemotherapy
  Proportion of patients with ototoxic hearing loss in total patients